CLINICAL TRIAL: NCT04781335
Title: "A Prospective Study of the Efficacy of Intracameral Dexamethasone (Dexycu™) Compared to Standard of Care Treatment for Post-Cataract Surgical Pain and Anterior Chamber Inflammation"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Eye Institute of West Florida (Other)
Collaborators: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EIWF-EP001
Record Dates: First submitted 2021-02-12; First posted 2021-03-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cataract
Keywords: Cataract; Dexycu
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate; Steroids; Anti-Bacterial Agents; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexycu (Active Comparator)
  Interventions: Drug: Dexycu
- Standard Care Post operative drops (Active Comparator)
  Interventions: Drug: Standard of Care post operative eye drops (steroid, antibiotic, NSAID)

INTERVENTIONS:
Drug: Dexycu — This is a contra-lateral randomized study, meaning that in clinic after a patient is identified as a candidate we will "flip a coin" for selection of the eye that is going to receive the Dexycu™ implant (the implant will be placed intracapsularly at the optic haptic junction of the IOL). The patients will receive the SAME topical regimen (Eye with Dexycu™: no steroid, Eye without Dexycu™: steroid will be used). The Dexycu™, topical NSAID, and antibiotic regimen will be provided to all patients in the study, at no cost, in order to avoid difficulties with compliance, insurance, and follow up.
  Arms: Dexycu
Drug: Standard of Care post operative eye drops (steroid, antibiotic, NSAID) — This is a contra-lateral randomized study, meaning that in clinic after a patient is identified as a candidate we will "flip a coin" for selection of the eye that is going to receive the Dexycu™ implant (the implant will be placed intracapsularly at the optic haptic junction of the IOL). The patients will receive the SAME topical regimen (Eye with Dexycu™: no steroid, Eye without Dexycu™: steroid will be used). The Dexycu™, topical NSAID, and antibiotic regimen will be provided to all patients in the study, at no cost, in order to avoid difficulties with compliance, insurance, and follow up.
  Arms: Standard Care Post operative drops

SUMMARY:
Cataract surgery is the most common surgical procedure performed on humans today. The postoperative regimen includes a combination of steroids, NSAIDs (non-steroidal anti-inflammatory drugs) and antibiotics. Those are used to decrease the possibility of infection, inflammation that may lead to corneal and macular edema and pain management. There are several FDA approved agents either for topical use as single drug delivery or combination solutions for topical use as well; furthermore, there are slow release vehicles that may be placed at the time of surgery or postoperatively (at the lower punctum). The latter provides a less intense and demanding drop schedule and may improve patient compliance.

DETAILED DESCRIPTION:
The current study will assess post cataract the efficacy and safety of two different FDA approved regimens, which include the standard of care (topical steroids, NSAIDs and antibiotics) or Intracameral Dexamethasone (Dexycu™) along with topical NSAIDs and antibiotics.

The hypothesis of the current study is that topical steroids or intracamerally injected steroids as slow release vehicles, demonstrate the same efficacy of controlling post cataract pain and inflammation. We will assess one objective outcome measure, anterior chamber inflammation. This will provide a direct index of the efficacy of the steroidal agents used. Furthermore, a subjective outcome measure, ocular pain, will also be assessed. In cases where a patient in either of the two groups has sever inflammation, rescue medications will be applied, increasing the dosage of topical steroidal agents and the patient will be followed closely until resolved.

The study will include 50 consecutive patients, men and women ages 40 to 90 years old, with visually significant cataract that received bilateral cataract surgery using either the manual technique or femtosecond assisted cataract surgery. Bilateral surgery is common practice and is not performed on the same day. There is a one week time interval between the eyes receiving cataract extraction. The patients that we will enroll in the suggested study will require and will receive bilateral cataract surgery with one week time interval between the two eyes. There are no restrictions on racial or ethnic origin. Employees of The Eye Institute of West Florida will not be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* • Patients age 40 to 90 years old, with visually significant cataract that received bilateral cataract surgery using either the manual technique or femtosecond assisted cataract surgery

Exclusion Criteria:

* • Patients with history of diabetes mellitus and other systemic conditions that may promote inflammation

  * patients with previous ocular disease history
  * patients with history of ocular surgery
  * patients using prescription eye medications topically
  * vulnerable subjects or subjects with diminished capacity requiring a POA (Power of Attorney)
  * patients with allergies to steroids, NSAID's, or besifloxacin (standard antibiotic)
  * women who are pregnant or lactating

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Pain score | post operative day 1
  Concerning the outcome measures of pain we are going to use NRS pain (numeric rating scale score) that takes a minute to do, it is a subjective measure of pain that the patient is experiencing, the patient circles a number between 0 and 10 (0 no pain and 10 worse pain imaginable). Score 0 will be considered as no pain and any score equal or more than 5 will be considered as moderate to severe pain.
Pain score | post operative day 7
  Concerning the outcome measures of pain we are going to use NRS pain (numeric rating scale score) that takes a minute to do, it is a subjective measure of pain that the patient is experiencing, the patient circles a number between 0 and 10 (0 no pain and 10 worse pain imaginable). Score 0 will be considered as no pain and any score equal or more than 5 will be considered as moderate to severe pain.
Pain score | post operative day 30
  Concerning the outcome measures of pain we are going to use NRS pain (numeric rating scale score) that takes a minute to do, it is a subjective measure of pain that the patient is experiencing, the patient circles a number between 0 and 10 (0 no pain and 10 worse pain imaginable). Score 0 will be considered as no pain and any score equal or more than 5 will be considered as moderate to severe pain.
Inflammation Score | post operative day 1
  Concerning the outcome measures of cell and flare we are going to use SOIS (summed ocular inflammation score).
Inflammation Score | post operative day 7
  Concerning the outcome measures of cell and flare we are going to use SOIS (summed ocular inflammation score).
Inflammation Score | post operative day 30
  Concerning the outcome measures of cell and flare we are going to use SOIS (summed ocular inflammation score).

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Weinstock, MD, Principal Investigator — The Eye Institute of West Florida
Locations (1):
- The Eye Institute of West Florida, Largo, Florida, United States

IPD SHARING:
Plan to Share IPD: No